CLINICAL TRIAL: NCT01457196
Title: Development of a Tumor Molecular Analyses Program and Its Use to Support Treatment Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1108
Record Dates: First submitted 2011-10-13; First posted 2011-10-21 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Neoplasm
Keywords: Cancer Genetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sequencing Arm (Other)
  Interventions: Diagnostic Test: Tumor Genetic Sequencing

INTERVENTIONS:
Diagnostic Test: Tumor Genetic Sequencing — This study will look at genetic material from a sample of the subjects tumor, look at certain changes in the genetic material, and see if these changes are related to the subjects cancer.

SUMMARY:
The primary objective of this specimen correlative study is two-fold: to provide a mechanism for the association of known molecular alterations with clinical outcomes, and to provide rapid genetic profiling of alterations with known clinical utility using tumor and germline specimens to support treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Current or prospective cancer patients; current cancer patients must have histologically or cytologically confirmed diagnosis of cancer
2. Tumor tissue available and suitable for molecular analyses from at least one of the following sources:

   * Tissue previously stored in UNC's Tissue Procurement Facility (TPF)
   * Tissue previous stored at an institution other than UNC-CH, provided investigators can determine that the tumors were sampled and stored under appropriate conditions for inclusion in the study
   * Patient undergoing tissue collection as per clinical standard of care and willing to allow specimens from surplus tissue to be diverted for research purposes
   * Patient undergoing tissue collection as per clinical standard of care and willing to have additional specimens taken for research
   * Patient willing to undergo biopsy for purpose of research only
3. The following inclusion criteria apply only to patients undergoing biopsy for research purposes only under this protocol:

   * ≥18 years of age
   * Treatment options offer no expectation of cure, e.g., advanced solid tumor patients with metastatic disease. NOTE: This restriction applies to biopsy of vital organs only, e.g., lung, liver, etc.
   * Appropriate candidate for research biopsy based on institutional standards for target biopsy site

Exclusion Criteria:

1. Any condition that would make participation in the protocol unreasonably hazardous for the patient in the opinion of the treating physician
2. Dementia, altered mental status, or any psychiatric condition or co-morbid condition that would prohibit the understanding or rendering of informed consent.
3. The following exclusion criteria apply only to enrolled patients undergoing biopsy for research purposes only:
4. History of serious or life-threatening allergic reaction to local anesthetics (i.e. lidocaine, xylocaine) or any medications used for conscious sedation (if applicable).
5. Requires general anesthesia for collection of biopsy
6. Pregnant or lactating women
7. Active cardiac disease
8. Patients receiving bevacizumab less than 6 weeks prior to enrollment into this study should not undergo research core biopsies because of the concern for potential increased bleeding risk and delayed healing. (NOTE: Patients receiving bevacizumab who are undergoing a research biopsy of accessible organs (e.g. breast, lymph node, skin etc.) must be two weeks from the last dose of the angiogenesis inhibitor).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2798 (Actual)
Dates: Start 2011-09; Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Shelton Earp, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 2798 participants screened for eligibility, 2074 were deemed eligible, 459 failed processing/sequencing, 226 had a sample collection failure, 19 were pediatric patients who were excluded from the final cohort, and 20 consents were withdrawn.
Groups:
- Sequencing Arm: All eligible subjects who had Tumor Genetic Sequencing performed. This sequencing looked at genetic material from a sample of the subjects tumor and certain changes in the genetic material, to see if these changes are related to the subjects cancer.
Period: Overall Study
Arm/Group | Sequencing Arm
Started | 2074
Completed | 2074
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sequencing Arm
Number analyzed (Participants) | 2074
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1482
  >=65 years | 592
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1352
  Male | 722
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67
  Not Hispanic or Latino | 1972
  Unknown or Not Reported | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 327
  White | 1573
  More than one race | 3
  Unknown or Not Reported | 125
Region of Enrollment [Number; unit: participants]
  United States | 2074

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Reportable Genetic Variant
Description: To estimate the proportion of patients enrolled on the study who have undergone successful sequencing and have a reportable genetic variant identified
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Sequencing Arm
Number analyzed (Participants) | 2074
proportion of participants | 0.61 [0.59 to 0.63]

2. Primary Outcome: Progression Free Survival
Description: Estimate Progression Free Survival (PFS) at 2 years in cancer patients with active disease with a reportable genetic variant and those without a reportable genetic variant
Time Frame: 2 Year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Reported: Subjects with next-generation sequencing who had somatic variants identified by the University of North Carolina (UNC )Molecular Tumor Board as actionable that were unknown at the time of testing reported to their treating physicians.
- Not Reported: Subjects with next-generation sequencing who had no somatic variants identified by the UNC Molecular Tumor Board as actionable that were unknown at the time of testing reported to their treating physicians.
Arm/Group | Reported | Not Reported
Number analyzed (Participants) | 1267 | 807
percentage of participants | 31 [26 to 37] | 62 [53 to 70]

3. Other Pre Specified Outcome: Collect and Describe Clinical Data
Description: To collect and describe clinical data including treatment outcomes after availability of results in patients
Time Frame: 1 Year
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Progression Free Survival
Description: To compare progression free survival ratios between cancer patients with active disease with reportable genetic variant who were treated based on variant and those who were not treated based on a variant
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Sequencing Arm
All-Cause Mortality (participants affected / at risk) | 723/2074
Serious Adverse Events (participants affected / at risk) | 0/2074
Other Adverse Events (participants affected / at risk) | 0/2074

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT01457196/Prot_SAP_000.pdf